CLINICAL TRIAL: NCT00725608
Title: Evaluation of Transfer From Subutex or Other Treatment for Opioid Drug Dependence to Suboxone: Acceptability, Safety and Impact on Medication Dispensing
Brief Title: Acceptability and Safety of Switching From Subutex or Other Opioid Drug Dependence Therapy to Suboxone (NIS P05444)
Status: Completed | Type: Observational
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P05444
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2012-03-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Opioid-Related Disorders; Opiate Dependence; Drug Abuse
Keywords: Suboxone; Subutex; Buprenorphine; Naloxone
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Opioid dependent patients currently in maintenance treatment with another medication who are switched to Suboxone (buprenorphine plus naloxone)
  Interventions: Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: buprenorphine/naloxone — 2/0.5 mg buprenorphine/naloxone and 8/2 mg buprenorphine/naloxone sublingual tablets; dosage and frequency are subject specific; subjects will receive treatment for up to 12 months
  Other Names: Suboxone, SCH 000484

SUMMARY:
The purpose of this study is to evaluate the acceptability and safety of switching to Suboxone® (buprenorphine plus naloxone) and the effect of the switch on medication dispensing. Subjects, for whom a therapy with Suboxone® is indicated and planned prior to study enrollment and who are willing to participate, will initiate therapy on Day 1 of the study. The dosage will be adjusted between Day 2 to 7 depending on patient's needs and determined by the treating physicians in accordance with the SmPC of Suboxone®. Data will be collected at baseline, day 1 til 7, the end of weeks 2 and 4 and monthly up to the end of Month 12.

DETAILED DESCRIPTION:
Nonprobability sampling was done by invitation to volunteer.

ELIGIBILITY:
Inclusion Criteria:

* All patients on substitution therapy, that are willing to switch to Suboxone, can be included.
* Therapeutic indications and contraindications for Suboxone® must be taken into consideration when selecting patients.

Exclusion Criteria:

* According to product information
* In accordance with the product information pregnant women will be excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients on substitution therapy for opioid dependence willing to switch to Suboxone
Sampling Method: Non-Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2008-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fischer, Prof. Dr., Principal Investigator — Medical University Vienna
Locations (1):
- (Multiple sites in Austria) => Coordinating CRO: H&P GmbH, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: May 2008 - December 2009 Patients were eligible for observation if the transfer from an ongoing opioid dependence therapy to Suboxone was indicated and planned prior to enrollment to P05444 by the treating physician.
  Multiple sites in Austria: general practitioners, clinics/outpatient clinics, drug counseling centers, prisons
Pre-assignment Details: 339 patients were enrolled, 32 datasets were excluded from analysis because of missing baseline assessment and/or missing final/dropout documentation = 307 eligible datasets were used for final general and safety analysis
Groups:
- Opioid Dependent Patients: Opioid dependent patients currently in maintenance treatment with another medication who are switched to Suboxone (buprenorphine plus naloxone)
Period: Overall Study
Arm/Group | Opioid Dependent Patients
Started | 307 (339 patients enrolled, 32 non-eligible datasets excluded from final general and safety analysis)
Completed | 140 (1 patient terminated treatment at day 368 and was counted as dropout)
Not Completed | 167
Not completed — Lost to Follow-up | 60
Not completed — Adverse Event | 14
Not completed — Individual reasons | 86
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Arm/Group | Opioid Dependent Patients
Number analyzed (Participants) | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.3 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 234
Region of Enrollment [Number; unit: participants]
  Austria | 307

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate
Description: The primary objective of this study was to determine the retention rate of patients after 6 and 12 months of treatment with buprenorphine/naloxone measured by the percentage of patients remaining in the study
Time Frame: month 6, month 12
Population: All eligible datasets were included in analysis population.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Opioid Dependent Patients
Number analyzed (Participants) | 307
percentage of patients
  Retention rate after 6 months of treatment | 57.3 [51.8 to 62.9]
  Retention rate after 12 months of treatment | 45.6 [40.0 to 51.2]

2. Secondary Outcome: Dosing of Suboxone (Buprenorphine Plus Naloxone)
Description: One of the secondary objectives was to evaluate the effect of the switch to buprenorphine/naloxone on medication dispensing measured by dose.
Time Frame: day 1, month 6, month 12
Population: All participants with eligible datasets were included in the final analysis
Measure: Mean (Standard Deviation); unit: Dose of Suboxone® in mg
Arm/Group | Opioid Dependent Patients
Number analyzed (Participants) | 307
Dose of Suboxone® in mg
  Suboxone® dose day 1 (mg) | 7.7 (4.9)
  Suboxone® dose month 6 (mg) | 9.1 (5.1)
  Suboxone® dose month 12 (mg) | 8.5 (4.8)

3. Secondary Outcome: Dispensing of Suboxone (Buprenorphine Plus Naloxone)
Description: Another of the secondary objectives was to evaluate the effect of the switch to Suboxone (buprenorphine plus naloxone) on medication dispensing measured by frequency of visits to the treating physician or pharmacy to receive the medication (daily, biweekly, once weekly, monthly, other)
Time Frame: month 6, month 12
Population: All participants with eligible datasets were included in the final analysis
Measure: Number; unit: Participants
Arm/Group | Opioid Dependent Patients
Number analyzed (Participants) | 307
Participants
  N patients with dispensing data at month 6 | 183
  6 month: Daily | 96
  Month 6: Biweekly | 1
  Month 6: Once weekly | 79
  Month 6: Monthly | 2
  Month 6: Other | 5
  N patients with dispensing data at month 12 | 142
  Month 12: Daily | 68
  Month 12: Biweekly | 1
  Month 12: Once weekly | 63
  Month 12: Monthly | 1
  Month 12: Other | 9

ADVERSE EVENTS:
Time Frame: Adverse events were collected for total observational time of each patient: from start of treatment until end of observation or date of early discontinuation, respectively - maximum period 1 year
Description: For description of safety data all patients enrolled and exposed to Suboxone® for at least one day(N=339) were included in the safety analysis
Arm/Group | Opioid Dependent Patients
Serious Adverse Events (participants affected / at risk) | 2/339
Other Adverse Events (participants affected / at risk) | 49/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid Dependent Patients (N=339)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) — Hospitalization
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) — no further information available
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid Dependent Patients (N=339)
Gastrointestinal disorders (Gastrointestinal disorders) | 25 (43)
General disorders and administration site conditions (General disorders) | 24 (36)
Psychiatric disorders (Psychiatric disorders) | 17 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results belong to the Sponsor only, all investigators are not allowed to publish study results without permission of the Sponsor.